CLINICAL TRIAL: NCT06070818
Title: Healthy Body & Mind Program: A Pilot Randomised Controlled Trial to Improve Quality of Life, Reduce Pain, and Reduce Dementia Risk in People Living With Cognitive Decline and Osteoarthritis
Brief Title: Healthy Body & Mind Program for Older Adults Living With Osteoarthritis and Cognitive Decline
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Claire Burley, Principal Investigator Dr Claire Burley, The University of New South Wales
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HC230506
Record Dates: First submitted 2023-09-25; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Cognitive Decline; Osteoarthritis
Keywords: dementia; lifestyle; multidisciplinary; physical activity; nutrition; depression; anxiety; pain; osteoarthritis; cognitive decline
MeSH Terms: conditions — Cognitive Dysfunction; Osteoarthritis; Dementia; Motor Activity; Depression; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: A randomised trial with a wait-list control.
Who Masked: Outcomes Assessor
Masking Description: The researcher collecting the outcome measures will not know whether the person is in the intervention or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Healthy Body & Mind Program: In summary, the program includes two visits to the University of New South Wales (UNSW) Medicine & Health Lifestyle Clinic at the beginning and end of the program for Initial and Final Assessments, and two weekly sessions for 12 weeks (24 sessions in total) to the UNSW Medicine & Health Lifestyle Clinic to complete the Healthy Body & Mind Program. Participants will also be invited to take part in a focus group either at the clinic or online (via Teams/ zoom) at the end of the program.
  Interventions: Other: Healthy Body & Mind Program
- Wait-list control (No Intervention): Usual care. Participants will not be recruited if they are taking part in another research intervention or receiving treatment other than usual care.

INTERVENTIONS:
Other: Healthy Body & Mind Program — 12-week physical activity and lifestyle education program
  Arms: Intervention

SUMMARY:
The goal of this pilot randomised clinical trial is to compare a 12-week Healthy Body & Mind Program to usual care in older adults living with cognitive decline and osteoarthritis.

The main questions it aims to answer are:

* Does the Healthy Body & Mind Program improve health-related quality of life in older adults living with cognitive decline and osteoarthritis (pre/post and intervention/control)?
* Does the Healthy Body & Mind Program improve other health outcomes (cognition, pain, anxiety/depression, physical function) in older adults living with cognitive decline and osteoarthritis (pre/post and intervention/control)?

Participants will complete a co-designed and multidisciplinary 12-week program that includes physical activity and lifestyle education (nutrition, social activity and managing anxiety/depression). Researchers will compare outcomes between the intervention group and a wait-list control to see if there are difference in outcome measures (quality of life, cognition, pain, anxiety/depression, physical function).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 55 or above.
* Montreal Cognitive Assessment score 18-25 indicating mild cognitive decline or mild dementia.
* Diagnosed with osteoarthritis.
* Able to safely undertake study assessments and complete exercise without assistance.

Exclusion Criteria:

* Montreal Cognitive Assessment score below 18.
* Display an abnormal cardiovascular response to exercise (as seen during the baseline exercise test) and your doctor does not provide medical clearance to exercise.
* Are unable to speak English and do not have a translator.
* Have orthopedic or neuromuscular limitations that prevent you from performing the exercise.
* Are deemed unsuitable for group exercise sessions following initial assessment by an Accredited Exercise Physiologist within the UNSW Lifestyle Clinic.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-06-26 (Estimated); Study Completion 2024-07-28 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life questionnaire | 12 weeks
  EuroQoL health-related quality of life (EQ-5D; https://euroqol.org/); Score range 0-1; 1 indicating full health, 0 indicating bad health.

SECONDARY OUTCOMES:
Cognition questionnaire | 12 weeks
  Montreal Cognitive Assessment (MoCA); Score range 0-30; higher scores mean better cognition. Measure can also be broken down into subscales.

OTHER OUTCOMES:
Chronic pain questionnaire | 12 weeks
  Western Ontario and McMaster Universities Arthritis Index (WOMAC); Score range 0-96; 0 represents best health, higher scores indicate more pain. Measure can also be broken down into subscales (e.g., pain and function).
Depression, anxiety & stress questionnaire | 12 weeks
  Depression Anxiety Stress Scales (DASS-21); Score range 0-21; higher scores mean worse psychological health. Measure can also be broken down into subscales: depression, anxiety & stress.
Physical function: 6-minute walk test | 12 weeks
  Assesses distance in metres walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance. Higher number of metres walked means better physical function and aerobic capacity.
Cardiovascular disease (CVD) risk profile questionnaire | 12 weeks
  ADCVD (https://tools.acc.org/ascvd-risk-estimator-plus/#!/calculate/estimate/). Tool calculated % risk, higher % indicates greater risk for CVD.
Sleep questionnaire | 12 weeks
  Pittsburgh Sleep Quality Index (PSQI); Score range 0-21; higher scores indicate worse sleep)
Physical function: handgrip strength physical test | 12 weeks
  Accesses physical strength in kilograms (kg). Average score of 3 attempts on each hand using a dynamometer; higher kg indicates more strength.
Physical function: single leg stance test (balance) physical test | 12 weeks
  Physical test used to assess static postural and balance control. The participant must stand unassisted on one leg and is timed in seconds from the time one foot is flexed off the floor to the time when it touches the ground or the standing leg or an arm leaves the hips. Higher number of seconds indicates better balance.

CONTACTS AND LOCATIONS:
Locations (1):
- UNSW Medicine & Health Lifestyle Clinic, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burley CV, Yeates W, McLeod KA, Jones MD, Borges N, Brodaty H, Parmenter BJ. Healthy Body and Mind Program to Improve Health Outcomes and Reduce Dementia Risk in People With Osteoarthritis: Protocol for a Feasibility and Acceptability Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Nov 6;14:e75816. doi: 10.2196/75816. PMID 41197122